CLINICAL TRIAL: NCT05031897
Title: A 2 Step Approach to Haploidentical Transplant Using Radiation-Based Reduced Intensity Conditioning
Brief Title: Two Step Haplo With Radiation Conditioning
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21D.466; JT 15545 (Other: JeffTrial Number)
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Adult T-Cell Leukemia/Lymphoma; Aplastic Anemia; Chronic Lymphocytic Leukemia; Chronic Myeloid Leukemia, BCR-ABL1 Positive; Chronic Myelomonocytic Leukemia; Essential Thrombocythemia; Hematopoietic and Lymphatic System Neoplasm; Hodgkin Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome; Myelofibrosis; Myeloid Neoplasm; Non-Hodgkin Lymphoma; Polycythemia Vera; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Aplastic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Thrombocythemia, Essential; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma, Non-Hodgkin; Polycythemia Vera | interventions — fludarabine; fludarabine phosphate; Whole-Body Irradiation; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Melphalan; Biopsy; X-Rays; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Radiation-Based Cohort (fludarabine, TBI, infusion) (Experimental): Patients receive fludarabine IV on days -11, -10, -9, and -8, undergo TBI BID on days -10 and -9, undergo DLI on day -6, and receive cyclophosphamide IV on days -3 and -2. Patients begin tacrolimus and mycophenolate mofetil IV on day -1. Patients then undergo HSCT on day 0. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy/aspiration, imaging and blood sample collection throughout the study.
  Interventions: Drug: Fludarabine; Radiation: Total-Body Irradiation; Procedure: Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Procedure: Hematopoietic Cell Transplantation; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Diagnostic Imaging; Procedure: Biospecimen Collection
- Arm 2: Chemotherapy-Based Cohort (fludarabine, melphalan, TBI) (Experimental): Patients receive fludarabine IV on days -11, -10, -9, and -8 and melphalan IV on days -10 and -9. Patients undergo TBI and DLI once on day -6. Patients receive cyclophosphamide IV on days -3 and -2 and begin tacrolimus and mycophenolate mofetil on day -1. Patients undergo hematopoietic stem cell transplant on day 0. Patients undergo bone marrow biopsy/aspiration, imaging and blood sample collection throughout the study.
  Interventions: Drug: Fludarabine; Radiation: Total-Body Irradiation; Procedure: Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Procedure: Hematopoietic Cell Transplantation; Drug: Melphalan; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Diagnostic Imaging; Procedure: Biospecimen Collection
- Arm 3: HLA- Identical cohort (radiation-based or chemotherapy-based conditioning) (Experimental): This group (HLA- Identical cohort), which is expected to be small, can undergo HSCT with radiation-based or chemotherapy-based conditioning. Due to small numbers of patients with available HLA identical related donors, this third, descriptive arm is included so that this group, too small in number for a free-standing study, are treated on clinical trial. This is also a separate arm of the study and the outcome of patients treated on this arm will be analyzed descriptively without statistical comparison or power analysis.
  Interventions: Drug: Fludarabine; Radiation: Total-Body Irradiation; Procedure: Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Procedure: Hematopoietic Cell Transplantation; Drug: Melphalan; Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Diagnostic Imaging; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine; 21679-14-1; 9-Beta-D-arabinofuranosyl-2-fluoro-9H-purin-6-amine; 9-Beta-D-arabinofuranosyl-2-fluoroadenine; Fluradosa
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; TOTAL BODY IRRADIATION; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
Procedure: Donor Lymphocyte Infusion — Undergo DLI
  Other Names: DLI; Donor Leukocyte Infusion
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 1-bis(2-chloroethyl)-amino-1-oxo-2-aza-5-oxaphosphoridin monohydrate; 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate; 2-[bis(b-chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane-2-oxide monohydrate; 2-[di(chloroethyl)amino]-1-oxa-3-aza-2-phosphacyclohexane 2-oxide monohydrate; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; 6055-19-2; Asta B 518; B 518; B-518; B518; bis(2-chloroethyl)phosphamide cyclic propanolamide ester monohydrate; Bis(2-chloroethyl)phosphoramide cyclic propanolamide ester monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; N,N-bis(2-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(2-chloroethyl)-N'-(3-hydroxypropyl)phosphorodiamidic acid intramolecular ester monohydrate, N,N-bis(2-chloroethyl)tetrahydro-2H-1,3,2-oxazaphosphorin-2-amine 2-oxide monohydrate; N,N-bis(b-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-propylenephosphoric acid ester diamide monohydrate; N,N-bis(beta-chloroethyl)-N',O-trimethylenephosphoric acid ester diamide monohydrate; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Tacrolimus — Given IV
  Other Names: 109581-93-3; FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Drug: Mycophenolate Mofetil — Given IV
  Other Names: 115007-34-6; 128794-94-5; Cellcept; MMF
Procedure: Hematopoietic Cell Transplantation — Undergo HSCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; HEMATOPOIETIC STEM CELL TRANSPLANT; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; NOS
Drug: Melphalan — Given IV
  Other Names: 148-82-3; 4-[bis(2-chloroethyl)amino]-L-phenylalanine; Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; p-di(chloroethyl)amino-L-phenylalanine; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Arm 2: Chemotherapy-Based Cohort (fludarabine, melphalan, TBI); Arm 3: HLA- Identical cohort (radiation-based or chemotherapy-based conditioning)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspiration/ biopsy
Procedure: Diagnostic Imaging — Undergo diagnostic imaging
  Other Names: Medical Imaging
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II clinical trial evaluates whether a modified modality of conditioning reduces treatment-related mortality (TRM) in patients who undergo a hematopoietic stem cell transplant (HSCT) for a hematological malignancy. HSCT is a curative therapy for many hematopoietic malignancies, however this regimen results in higher rates of TRM than other forms of treatment. In recent years, less intense conditioning regimens with radiation and chemotherapy prior to HSCT have been developed. Radiation therapy uses high energy sources to kill cancer cells and shrink tumors while chemotherapy drugs like fludarabine and cyclophosphamide work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This study evaluates whether a two-step approach with lower-intensity regimens of these treatments prior to HSCT reduces the rate of TRM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the 2 year cumulative incidence of TRM in patients undergoing reduced intensity conditioning (RIC) haploidentical (HI) HSCT in this protocol.

SECONDARY OBJECTIVES:

I. To assess the 2 year cumulative incidence of relapse in patients undergoing RIC HI HSCT in this protocol.

II. To assess the consistency and pace of engraftment. III. To assess the pace of T cell and B cell immune recovery. IV. To assess the incidence and severity of graft versus host disease (GVHD).

OUTLINE: Patients are assigned to 1 of 2 cohorts.

RADIATION-BASED COHORT: Patients receive fludarabine intravenously (IV) on days -11, -10, -9, and -8, undergo total-body irradiation (TBI) twice a day (BID) on days -10 and -9, undergo donor lymphocyte infusion (DLI) on day -6, and receive cyclophosphamide IV on days -3 and -2. Patients begin tacrolimus and mycophenolate mofetil IV on day -1. Patients then undergo HSCT on day 0. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy/aspiration, imaging and blood sample collection throughout the study.

CHEMOTHERAPY-BASED COHORT: Patients receive fludarabine IV on days -11, -10, -9, and -8 and melphalan IV on days -10 and -9. Patients undergo TBI and DLI once on day -6. Patients receive cyclophosphamide IV on days -3 and -2 and begin tacrolimus and mycophenolate mofetil on day -1. Patients undergo HSCT on day 0. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy/aspiration, imaging and blood sample collection throughout the study.

After completion of study treatment, patients are followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Radiation-based cohort diagnoses:

  * Acute myeloid leukemia
  * Acute lymphoid leukemia in remission
  * Myelodysplasia (MDS)
  * Chronic lymphocytic leukemia (CLL) with no or minimal lymph node involvement
  * Multiple myeloma
  * Chronic myeloid leukemia
  * Myelofibrosis
  * Myeloid malignancy not otherwise specified
  * Chronic myelomonocytic leukemia
  * Essential thrombocytopenia or polycythemia vera
  * T cell leukemia
  * T cell lymphoma without significant lymph node disease burden
  * Any hematological malignancy or dyscrasia not cited above in which HSCT is potentially curable
  * Any patient who has a hematological disease that would normally be treated on a myeloablative study, but is prevented from doing so by factors in their past medical history. Examples are patients with previous treatment with radiation therapy precluding total-body irradiation (TBI), or a past history of myeloablative therapy, precluding a 2nd myeloablative regimen.
  * Patients must have a donor who is one-haplotype mismatched (number of mismatches in either direction not considered)
* Chemotherapy-based cohort diagnoses:

  * Hodgkin or non-Hodgkin lymphoma
  * Small lymphocytic lymphoma/CLL
  * Any other diagnosis in which chemotherapy is thought to be superior to radiotherapy for treatment of the disease
  * Hematological malignancy in patients who cannot receive > 2 Gy radiation
  * Aplastic anemia and other non-malignant hematologic dyscrasias
  * Patients must have a donor who is one-haplotype mismatched (number of mismatches in either direction not considered)
* Human leukocyte antigen (HLA) identical cohort diagnoses:

  * Patients in this group will be treated in parallel to the radiation-based cohort or the chemotherapy-based group based on what category their diagnosis falls into. However, these patients will have HLA identical related donors (one-antigen cross-over event included).
* Left ventricular ejection fraction of >= 50%
* Diffusion lung capacity of oxygen >= 50% and forced expiratory volume at 1 second >= 50% of predicted corrected for hemoglobin
* Serum bilirubin =< 1.8
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x upper limit of normal
* Creatinine clearance of >= 60 mL/min
* Patients must have adequate Karnofsky performance status (KPS) and Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) scores:

  * Patients < age 60 years must have a KPS of >= 60% and an HCT-CI score of 5 or less
  * Patients aged 60 to 65 years must have a KPS of >= 60% and an HCT-CI score of 4 or less
  * Patients aged 66 to 69 years must have a KPS of 90% and an HCT-CI score of 3 or less
  * Patients aged 70 years or more must have a KPS of 90% and an HCT-CI score of 2 or less
  * (Patients with greater than the allowable HCT-CI points for age can be enrolled for trial with approval of the principal investigator (PI) and at least 1 co-investigator (CI) not on the primary care team of the patient). This is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than guideline HCT-CI points. An example is a patient with a solid tumor malignancy in their remote history (adds 3 points to HCT-CI total) where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities
* Patients must be willing to use contraception if they have childbearing potential
* Patient or patient's guardian is able to give informed consent
* Patients should have a life expectancy of >= 6 months for reasons other than their underlying hematologic/oncologic disorder
* Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol
* Patients should not be:

  * Human immunodeficiency virus positive
  * Have active involvement of the central nervous system with malignancy. This can be documented by a normal neurological exam, magnetic resonance imaging (MRI) of the head, and/or a negative cerebral spinal fluid analysis
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience Treatment-Related Mortality (TRM) | At 2 years post hematopoietic stem cell transplant (HSCT)
  TRM is defined as death without evidence of recurrent disease in the 2 year period post HSCT. Summarized using Kaplan-Meier curves and the respective Kaplan-Meier estimates of the 2-year event rate are reported as well as their 95% confidence intervals.

SECONDARY OUTCOMES:
Development of relapsed disease | Up to 2 years
  Relapse is measured by evidence of recurrent disease in the blood, marrow, or lymph nodes. Summarized using Kaplan-Meier curves and the respective Kaplan-Meier estimates of the 2-year event rate are reported as well as their 95% confidence intervals.
Engraftment | Up to 2 years
  Measure by chimerism studies of the blood and marrow at multiple time points after the HSCT. Chimerism refers to the percentage of donor cells in the hematopoietic system of the patient post HSCT. Reported using mean and standard deviations.
Immune reconstitution | Up to 2 years
  Evaluated by T-cell recovery and B-cell recovery. Assessed by the quantitative measurement of CD3/4 and CD3/8 cells and immunoglobulin levels in the blood at multiple time points post HSCT. CD3/4 and CD3/8 counts are measured by an immune reconstitution panel and immunoglobulin levels are measured by a quantitative immunoglobulin assay. Reported using mean and standard deviations
Incidence and degree of graft versus host disease (GVHD) after HSCT | Up to 2 years
  Assessment includes presence and degree of skin rash, presence and amount of diarrhea, and/or abnormal liver function test. Summarized using Kaplan-Meier curves and the respective Kaplan-Meier estimates of the 2-year event rate are reported as well as their 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Usama Gergis, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadephia, Pennsylvania, United States